CLINICAL TRIAL: NCT07161271
Title: Retrospective Cohort Study of Low-Flow Extracorporeal Carbon Dioxide Removal (ECCO2R) System: Evaluating Efficacy and Safety
Brief Title: Retrospective Cohort Study of Low-Flow Extracorporeal Carbon Dioxide Removal (ECCO2R) System: Evaluating ECCO2R's Efficacy and Safety in Participants With Respiratory Failure
Status: Recruiting | Type: Observational
Sponsor: Hong Kong University (Other)
Responsible Party: Principal Investigator, Simon Sin Wai-ching, Doctor; Director and Clinical Associate Professor, Hospital Authority, Hong Kong
Other Study IDs: UW 24-480; HKU/HA HKW IRB (Other: HKU/HA HKW Institutional Review Board)
Record Dates: First submitted 2025-08-20; First posted 2025-09-08 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-08

CONDITIONS: Respiratory Failure; ICU; Asthma (Diagnosis); ARDS
Keywords: ECCO2R; ICU; Asthma; ARDS; Respiratory failure
MeSH Terms: conditions — Respiratory Insufficiency; Asthma; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with respiratory failure and supported with ECCO2R: Patients supported with ECCO2R in one of the designated study sites; Admitted to the ICU between 1 Jan 2022 and 30 June 2024; Patients older than 18 years old

SUMMARY:
This is an observational study performed by retrospective review of data routinely collected for patients receiving low-flow extracorporeal carbon dioxide removal (ECCO2R) therapy in intensive care units (ICUs). Our aim is to firstly, describe the local practice in terms of patient selection and technical details of clinical management related to the use of low-flow ECCO2R system, and secondly, the clinical results in terms of patient outcomes and adverse events. These findings may allow clinicians to improve the quality and safety of ECCO2R therapy provision in the ICU.

DETAILED DESCRIPTION:
Extracorporeal carbon dioxide removal (ECCO2R) is a specialised medical procedure employed to eliminate excessive carbon dioxide (CO2) from the bloodstream. To date, there have been only a few small-scale studies published on ECCO2R, with limited data on the full spectrum of clinical presentations, management strategies, and outcomes. Previous clinical trials have investigated the potential for ECCO2R therapy to reduce the intensity of mechanical ventilation in patients suffering from acute respiratory distress syndrome (ARDS). While these trials have successfully achieved desired physiological outcomes, they have not consistently translated into improved patient mortality rates. Additionally, the use of ECCO2R has presented certain complications, especially when higher-flow ECCO2R systems based on the centrifugal pump technology were used, which had been more extensively studied in the past. However, our clinical experience appeared to suggest that low-flow ECCO2R therapy could be managed with reasonable treatment success rate and limited complications. The investigators hypothesise that the use of low-flow ECCO2R therapy is clinically effective and safe for a selected group of ICU patients with acute respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients supported with ECCO2R in one of the designated study sites
* Admitted to the ICU between 1 Jan 2022 and 30 June 2024

Exclusion Criteria:

* Patients younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients supported with ECCO2R in our designated study sites
Sampling Method: Non-Probability Sample
Enrollment: 59 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Around 60 participants with respiratory failure as assessed for their clinical characteristics and outcomes | From November 2024 to September 2026 (Anticipated)
  The primary endpoint is to describe the patients' demographics (e.g. Age, Sex), clinical characteristics (e.g. APACHE score, ventilator using time, respiratory parameters, ventilatory parameters, Mortality), outcomes of patients (death or survive) who received ECCO2R therapy.
  The secondary endpoints are to evaluate the association between clinical factors and patient outcomes (e.g. life of stay in ICU, ventilator free days), and to identify potential risk factors for adverse events and complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital (QMH), Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McNamee JJ, Gillies MA, Barrett NA, Perkins GD, Tunnicliffe W, Young D, Bentley A, Harrison DA, Brodie D, Boyle AJ, Millar JE, Szakmany T, Bannard-Smith J, Tully RP, Agus A, McDowell C, Jackson C, McAuley DF; REST Investigators. Effect of Lower Tidal Volume Ventilation Facilitated by Extracorporeal Carbon Dioxide Removal vs Standard Care Ventilation on 90-Day Mortality in Patients With Acute Hypoxemic Respiratory Failure: The REST Randomized Clinical Trial. JAMA. 2021 Sep 21;326(11):1013-1023. doi: 10.1001/jama.2021.13374. PMID 34463700
- [Result] Brodie D, Slutsky AS, Combes A. Extracorporeal Life Support for Adults With Respiratory Failure and Related Indications: A Review. JAMA. 2019 Aug 13;322(6):557-568. doi: 10.1001/jama.2019.9302. PMID 31408142
- [Result] Barbic B, Bianchi C, Madotto F, Sklar MC, Karagiannidis C, Fan E, Brochard L. The Failure of Extracorporeal Carbon Dioxide Removal May Be a Failure of Technology. Am J Respir Crit Care Med. 2024 Apr 1;209(7):884-887. doi: 10.1164/rccm.202309-1628LE. No abstract available. PMID 38190699
- [Result] Giraud R, Banfi C, Assouline B, De Charriere A, Cecconi M, Bendjelid K. The use of extracorporeal CO2 removal in acute respiratory failure. Ann Intensive Care. 2021 Mar 11;11(1):43. doi: 10.1186/s13613-021-00824-6. PMID 33709318
- [Result] Zhou Z, Li Z, Liu C, Wang F, Zhang L, Fu P. Extracorporeal carbon dioxide removal for patients with acute respiratory failure: a systematic review and meta-analysis. Ann Med. 2023 Dec;55(1):746-759. doi: 10.1080/07853890.2023.2172606. PMID 36856550
- [Result] Morelli A, Del Sorbo L, Pesenti A, Ranieri VM, Fan E. Extracorporeal carbon dioxide removal (ECCO2R) in patients with acute respiratory failure. Intensive Care Med. 2017 Apr;43(4):519-530. doi: 10.1007/s00134-016-4673-0. Epub 2017 Jan 28. PMID 28132075